CLINICAL TRIAL: NCT01096004
Title: A Randomised, Single-blind, Placebo-controlled, Single-centre, Phase I Study in Abdominally Obese Healthy Volunteers to Evaluate Methods to Assess 11-βHSD1 Activity in Adipose Tissue and Related Downstream Biomarkers After Single and Repeated Oral Doses of AZD4017 for 10 Days
Brief Title: Study to Evaluate Methods That Assess the Effect of AZD4017 in Adipose Tissue
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: D2060M00001
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Obesity
Keywords: Pharmacodynamic method evaluation
MeSH Terms: conditions — Obesity | interventions — 2-(1-(5-(cyclohexylcarbamoyl)-6-propylsulfanylpyridin-2-yl)-3-piperidyl)acetic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD4017
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD4017 — oral suspension, 1200mg, once daily, for 10 days
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The primary purpose of this study is to investigate different methods to evaluate the effect of AZD4017 in adipose tissue after single and multiple doses of AZD4017 in abdominally obese but otherwise healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written and dated informed consent
* Have a body mass index (BMI) between 27 and 35 kg/m2
* Waist circumference of >102 cm

Exclusion Criteria:

* History of any clinical significant disease
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of investigational product
* Any clinically significant abnormalities in clinical chemistry, haematology or urinalysis results as judged by the investigator

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of single and repeated doses of AZD4017 and placebo on mechanisms in adipose tissue involved in metabolic regulation | A adipose tissue biospy is taken at baseline, on first day of dosing day, on 4th dosing day and on 9th dosing day.

SECONDARY OUTCOMES:
Safety and Tolerability (Adverse events, vital signs, ECGs, physical examination, laboratory variables | The variables will be measure predose and the repeatedly during the following 10 days after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Per-Anders Jansson, Ass Prof, MD, PhD, Principal Investigator — Avdelningen för molekylär och klinisk medicin Lundberglaboratoriet; Mikaela Sjöstrand, Study Chair — AstraZeneca
Locations (1):
- Research Site, Gothenburg, Sweden